CLINICAL TRIAL: NCT06365996
Title: Development and Validation of the Polish Version of the Geriatric Categorical Profile Based on ICF.
Brief Title: Development and Validation of the Polish Geriatric Core Set.
Status: Not yet recruiting | Type: Observational
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Agnieszka Sozanska, dr hab. n. o zdr., prof. UR, University of Rzeszow
Other Study IDs: Core set geriatric ICF
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Aging
Keywords: aging, aged, ICF, disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Population ageing is a global problem. With ageing, involutionary changes and multimorbidity increase, leading to limitations in the performance of daily activities and disability. Proposed by the World Health Organisation (WHO), the geriatric core set is a set of categories of the International Classification of Functioning, Disability and Health (ICF) that allows for a comprehensive assessment of a person of geriatric age. In Poland, the geriatric core set has not yet been adapted and validated. Therefore, the aim of this study is the cultural adaptation and validation of the Polish version of the ICF-based categorical profile for the assessment of older people.

DETAILED DESCRIPTION:
Introduction: In Poland, as in many developed countries, the demographic structure of the population is changing due to the ageing of the population. As people grow older, involutionary changes intensify, and the often accompanying multimorbidity leads to deterioration in the functional capacity of the elderly. An additional problem for older people is reduced emotional state and reduced quality of life, as well as cognitive impairment. A very important element affecting the functioning of older people is their living environment, both physical and social. All these elements affect the functioning and disability of older people.

The World Health Organisation (WHO) has created the International Classification of Functioning, Disability and Health (ICF) based on a comprehensive biopsychosocial approach to the patient, on the basis of which WHO experts prepare categorical sets that allow a comprehensive assessment of people with different problems. One such set is the categorical profile (expanded and shortened version) prepared for the comprehensive assessment of older people (Geriatrics Comprehensive and Bref Core sets). The World Health Organisation encourages the use of the ICF and categorical profiles by all member countries. In Poland, this profile has not yet been adopted and validated.

The aim of this study is to culturally adapt and validate the Polish version of the ICF-based categorical profile for the assessment of older people. Mapping tools to the profile. Assessment of older people using the prepared tool.

Material and method: a minimum of 800 people aged 65 and over are planned to be included in the study. The project will be carried out in stages:

I preparation of the Polish version of the categorical profile for assessing older people and cultural adaptation of the tool. The cultural adaptation will consist of verifying the categories included in the categorical profile for assessing older people; II Mapping the tools/questions for assessing the different ICF categories included in the first version of the categorical profile.

III Conducting a survey using the tools mapped to the core set among older people in order to validate the constructed categorical profile and make the necessary adjustments to the toolkit and profile categories. The actual survey will be carried out by means of a face-to-face interview and a physical survey; IV Cross-sectional study conducted in the Podkarpackie Voivodeship to assess the health and functioning of older people using the prepared categorical profile with the mapped tools.

ELIGIBILITY:
Inclusion Criteria:

* age of respondents 60 years and older;
* informed and voluntary consent of the participant to participate in the study;
* cognitive condition enabling conducting a reliable interview regarding the current health situation and functioning of the subject.

Exclusion Criteria:

* age of respondents below 60 years;
* lack of participant's consent to participate in the study;
* severe cognitive impairment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly people aged 60 and over living in south-eastern Poland.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
ICF Geriatric core set | 2024-04/2024-12
  International Classification Functioning Disability and Health Geriatric core set comprehensive and short version

SECONDARY OUTCOMES:
Sociodemographic data of the sample | 2024-04/2024-12
  Sociodemographic data of the sample (eg.age, sex, education level, number of comorbidities, environmental factors)
Disability - WHODAS 2.0 v 36 item | 2024-04/2024-12
  The 36-item WHODAS 2.0 is used to measure general disability and disability in six domains:
  Do1 Cognition (6 items), Do2 Mobility (5 items), Do3 Self-care (4 items), Do4 Getting along (5 items), Do5 Life activities (8 items), and Do6 Participation (8 items). During the interview, the response refers to the last 30 days. Answers to the questions are rated on a 5-point scale identifying the level of di culty or problem (1 = none; 2 = mild; 3 = moderate; 4 = severe; 5 = extreme or cannot to do).

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Sozańska, prof, Principal Investigator — University of Rzeszow
Locations (1):
- University of Rzeszow, Rzeszów, Podkarpackie Voivodeship, Poland